CLINICAL TRIAL: NCT07261007
Title: Investigation of the Effectiveness of Flossing in Hemiplegic Patients With Shoulder Pain: Randomized Controlled Trial
Brief Title: Investigation of the Effectiveness of Flossing in Hemiplegic Patients With Shoulder Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Doç.Dr.Ömer Şevgin, Assoc.Prof.Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar76
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Shoulder Pain; Hemiplegia
MeSH Terms: conditions — Shoulder Pain; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): conventional physiotherapy
  Interventions: Other: control
- flossing group (Experimental): conventional physiotherapy + flossing
  Interventions: Other: flossing

INTERVENTIONS:
Other: control — conventional physiotherapy applications; TENS, hotpack, ultrasound and exercise.
  Arms: control
Other: flossing — conventional physiotherapy applications; TENS, hotpack, ultrasound and exercise.
  The floss band application will cover the area around the shoulder joint (specifically the deltoid, pectoralis major, and subscapularis). The bandage will be applied in a spiral pattern, starting from the mid-distal portion of the deltoid muscle and working distally to proximally. It will be applied with approximately 50% tension.
  Arms: flossing group

SUMMARY:
This study aims to contribute to clinical practice by investigating the effectiveness of flossband application on range of motion, functionality, pain and sleep quality in hemiplegic patients with shoulder pain.

DETAILED DESCRIPTION:
This study will be conducted at the NRL Physical Therapy Center. Participants must sign an informed consent form before starting the study. Participants will be randomly assigned to two groups: a control and an experimental group. A Visual Analog Scale will be used to assess pain. A score of 0 represents no pain, and a score of 10 represents unbearable pain. The Pittsburgh Sleep Quality Scale will be used to assess sleep quality. Assessments will be made before starting treatment and at the end of treatment after 6 weeks. The experimental group will receive conventional physical therapy and flossband application. This group will receive conventional physical therapy and flossband application three sessions per week, each session lasting approximately 40-50 minutes, for 6 weeks. The flossband application will cover the area around the shoulder joint (specifically the deltoid, pectoralis major, and subscapularis line). A spiral bandage will be applied starting from the mid-distal portion of the deltoid muscle, working distally from proximal to distal.

ELIGIBILITY:
Inclusion Criteria

* Individuals with a clinical diagnosis of stroke
* Individuals between the ages of 30 and 55
* Individuals experiencing hemiplegic shoulder pain (VAS ≥ 3) and/or limited joint movement
* Individuals who have been at least 6 months post-stroke (chronic phase)
* Individuals who have an active range of motion of at least 90° in shoulder flexion and abduction
* Individuals with stable vital signs
* Individuals who volunteer to participate in the study and who understand the purpose and process of the study and sign a written informed consent form

Exclusion Criteria

* Presence of serious orthopedic problems such as shoulder fractures, dislocations, or rotator cuff tears
* Presence of skin lesions or circulatory disorders that may prevent flossband application
* Spasticity in the affected arm (Modified Ashworth Scale ≥1)
* Those with a latex allergy to the flossband material
* Those with acute inflammatory conditions or acute pain

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index | 8 weeks
  It's a self-reported questionnaire consisting of two subgroups: pain and shoulder disability level. It consists of 13 questions: five for pain and eight for shoulder disability level. In the pain section, a visual analog scale score of 0 indicates no pain and 10 indicates the most severe pain. In the shoulder disability level section, a score of 0 indicates no difficulty and 10 indicates very difficult (I need help). Scoring is performed by measuring the distance between the individual's chosen point and 0 using a ruler and recording the score in centimeters. The total score is calculated by averaging the two subgroup scores. A higher score indicates shoulder pain and functional impairment.
The Pittsburgh Sleep Quality Index | 8 weeks
  Pittsburgh Sleep Quality Index; It evaluates sleep duration, sleep disturbance, sleep efficiency, subjective sleep quality, sleep medication use, daytime dysfunction, and sleep delay and consists of a total of 24 questions. 19 of them are self-report scales and 5 of them consist of questions to be answered by a friend or spouse. There are 7 components with 18 questions scored in the scale, and each component is evaluated between 0 and 3 points. The total score ranges from 0 to 21, and 5 or more is an indicator of "poor sleep quality".

CONTACTS AND LOCATIONS:
Overall Officials: Kübra UZUN, Study Chair — Uskudar University
Locations (1):
- Turkey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelly CF, Oliveri Z, Saladino J, Senatore J, Kamat A, Zarour J, Douris PC. The Acute Effect of Tissue Flossing on Pain, Function, and Perception of Movement: A Pilot Study. Int J Exerc Sci. 2023 Jul 1;16(3):855-865. doi: 10.70252/OKAO5505. eCollection 2023. PMID 37637031
- [Background] Chen J, Wang Q, Zhao Z, Song Q, Zhao P, Wang D. Acute effects of tissue flossing on boxers with chronic knee pain. Front Bioeng Biotechnol. 2025 Jan 14;12:1508054. doi: 10.3389/fbioe.2024.1508054. eCollection 2024. PMID 39877264
- [Background] Quiles-Sanchez LV, Baroutas I, Kyriakos G, Gravvanis N, Georgakopoulou VE, Trakas N, Damaskos C, Garmpi A, Garmpis N, Antoniou V, Farmaki P, Patsouras A, Voutyritsa E, Diamantis E. Medical Flossing and the Pilates Method: Their Effectiveness on the Strength, Endurance, and Functionality of Healthy Individuals. Cureus. 2021 Apr 29;13(4):e14758. doi: 10.7759/cureus.14758. PMID 34084682